CLINICAL TRIAL: NCT01302925
Title: PEP005 Gel - Evaluation of Local Tolerability After Exposure to Ingenol Mebutate 0.05% and 0.015% Gel Followed by Hand Washing in Healthy Subjects.
Brief Title: PEP005 Gel - Evaluation of Local Tolerability After Exposure to Ingenol Mebutate Gel Followed by Hand Washing in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peplin (Industry)
Collaborators: LEO Pharma (Industry)
Responsible Party: Rikke L Fischer/International Clinical Trial Manager, LEO Pharma
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: LP0041-01
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy; Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP005 Gel 0.05%/2 days (Experimental): Subjects will be exposed to investigational product for 2 consecutive days.
  Interventions: Drug: PEP005 Gel
- PEP005 Gel 0.015%/3 days (Experimental): Subjects will be exposed to investigational product for 3 consecutive days.
  Interventions: Drug: PEP005 Gel

INTERVENTIONS:
Drug: PEP005 Gel — PEP005 Gel 0.05% for 2 consecutive days
  Arms: PEP005 Gel 0.05%/2 days
Drug: PEP005 Gel — PEP005 Gel 0.015% for 3 consecutive days
  Arms: PEP005 Gel 0.015%/3 days

SUMMARY:
The purpose of this phase 1 trial is to investigate the local tolerability on the finger following exposure to PEP005 Gel 0.015% or 0.05% and hand washing once daily, for 2 or 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or female and at least 18 years of age
* Female patients must be of: non-childbearing potential or if of childbearing potential then have a negative serum and urine pregnancy test and using effective contraception
* Ability to provide informed consent

Exclusion Criteria:

* Have received treatment with immunomodulators, or interferon/interferon inducers or systematic medications that suppress the immune system in the last 4 weeks
* Exposed to prescribed systemic (take as tablet, injection etc) or topical (gel, cream, lotion) medication within the last 7 days
* Have any signs of skin irritation or damaged skin at or around the dominant index finger
* Have worked in an occupation with a high risk of being in contact with irritative material (eg. chemicals, painting) on their hands, especially fingers
* Those who are currently participating in any other clinical trial
* Those known or suspected of not being able to comply with the requirements of the protocol
* Females who are pregnant or are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Local Skin Responses | Up to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dosik, MD, Principal Investigator — TKL Research
Locations (1):
- TKL Research, Paramus, New Jersey, United States